CLINICAL TRIAL: NCT06075459
Title: Post Marketing Clinical Evaluation Assessing the Visual Performance of Hanita Lenses "Intensity SL" Intraocular Lens
Acronym: Post-op
Status: Completed | Type: Observational
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Other Study IDs: HTF-PM-AR
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cataract
Keywords: Cataract; IOL; Hanita Lenses
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Implanted patients with Intensity IOLs, 12-24 months previously: Men and women who had implantation on both eyes using Hanita Lenses SeeLens SL IOL, for 12 to 24 months post operation.

SUMMARY:
This clinical study will assess the safety and performance of Intensity SL IOL, 1 year post operation.

The study will also evaluate the patient satisfaction of the implanted patients.

DETAILED DESCRIPTION:
Study Design:

This study is an ambispective, single arm single center, open label study.

Study Objectives:

The aim of this study is to evaluate performance of Hanita Lenses Intensity SL IOL. The primary aim of this study is to evaluate the binocular defocus Curve and visual acuity for far, intermediate and near distance after Intensity SL IOL implantation.

The second aim of this study is to evaluate the patient satisfaction 12 to 24 months post-operation.

Study population:

Men and women who had implantation on both eyes using Hanita Lenses SeeLens SL IOL, for 12 to 24 months post operation.

Enrollment:

The study will encompass a total of 60 eligible subjects implanted bilaterally (120 eyes) in total who will complete the protocol follow-up schedule.

Duration of Subject participation:

Duration of Subject participation is at most one month Completion of active enrolment is anticipated to last approximately 6 months. The primary aim will be finally evaluated when the last study subject has been recruited.

Visits & Procedures Patients participating in the trial will attend a total of one visit (1 year follow up visit).

Subjects will be selected from the physician's usual subjects' practice. All subjects meeting the inclusion criteria and having signed the Informed Consent Form will be evaluated by the Investigator according to the study protocol.

1 year follow up visit: Pre-operation Visit: performed to check inclusion criteria, and to sign the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Implanted bilaterally using Hanita Intensity SL IOL
* 12 to 24 months post implantation
* Signed informed consent

Exclusion Criteria:

• Patients with any other pre-implantation and post implantation eye disease or condition that might affect the safety and efficacy evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women who had implantation on both eyes using Hanita Lenses SeeLens SL IOL, for 12 to 24 months post operation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to evaluate performance of Hanita Lenses Intensity SL IOL. | 21-24 months post operation
  Performance of the IOL will be evaluated by assessing the defocus Curve and visual acuity for far, intermediate and near distance after Intensity SL IOL implantation.

SECONDARY OUTCOMES:
The second aim of this study is to evaluate the patient satisfaction post-operation. | 21-24 months post operation
  Patient satisfaction will be evaluated by using Quality of Life (VH14) and satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: German Bianchi, MD, Principal Investigator — Dr. Nano Eye Clinic
Locations (1):
- Dr. Nano Eye Clinic, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No